CLINICAL TRIAL: NCT05508035
Title: The Effect of Sacubitril/valsartan Versus Ramipril on Left Ventricular Function and Remodeling in Patients with Ischemic Heart Failure with Mid-range Ejection Fraction
Acronym: CRACOVIA-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW.0701.005.2020P
Record Dates: First submitted 2022-08-11; First posted 2022-08-19 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure with Moderately Reduced Ejection Fraction
Keywords: chronic heart failure; congestive heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sacubitril / valsartan (Experimental): sacubitril / valsartan 200 mg twice a day PLUS placebo for ramipril 5 mg twice a day
  Interventions: Drug: Sacubitril / Valsartan
- ramipril (Active Comparator): ramipril 5 mg twice a day PLUS placebo for sacubitril / valsartan 200 mg twice a day
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Sacubitril / Valsartan — The participants will be randomized to either ramipril 5 mg twice daily plus placebo for sacubitril / valsartan 200 mg twice daily or sacubitril / valsartan 200 mg twice daily plus placebo for ramipril 5 mg twice daily in 1: 1 ratio using the IT randomization module. All patients eligible for randomization will receive their first dose of double-blind drug plus placebo the day after randomization visit. After assigning a randomized treatment, patients will continue at the target dose and attend a 2-week telephone follow-up followed by site visits after one month, four months, eight months and in the final visit after 12 months.
  Arms: sacubitril / valsartan
Drug: Ramipril — The participants will be randomized to either ramipril 5 mg twice daily plus placebo for sacubitril / valsartan 200 mg twice daily or sacubitril / valsartan 200 mg twice daily plus placebo for ramipril 5 mg twice daily in 1: 1 ratio using the IT randomization module. All patients eligible for randomization will receive their first dose of double-blind drug plus placebo the day after randomization visit. After assigning a randomized treatment, patients will continue at the target dose and attend a 2-week telephone follow-up followed by site visits after one month, four months, eight months and in the final visit after 12 months.
  Arms: ramipril

SUMMARY:
Heart failure with moderately reduced ejection fraction (HFmrEF) is a frequent disease associated with significant morbidity and mortality and therefore requires effective therapies that may improve clinical outcomes. The most common reason of HFmrEF is ischemic injury, usually caused by myocardial infarction, that may lead to left ventricular remodeling and systolic dysfunction, accompanied by symptoms of heart failure. Therefore, the anti-remodeling therapies may effectively improve clinical outcomes. Recently, sacubitril/valsartan - the angiotensin receptor neprilysin inhibitor suppressing the renin-angiotensin-aldosterone system and enhancing the effect of natriuretic peptides - has been introduced in the treatment of heart failure. To date, this drug was found to be clinically beneficial in patients with heart failure with reduced ejection fraction (HFrEF), however has not been tested in the group of patients with HFmrEF.

The aim of the study is to evaluate effectiveness of sacubitril/valsartan as compared with ramipril on left ventricular remodeling and function in patients with ischemic HFmrEF.

Patients with ischemic HFmrEF, New York Heart Association class II-IV symptoms, an elevated plasma natriuretic peptide level and the left ventricular ejection fraction (LVEF) of 40-49 % will be enrolled in this prospective, multicenter, randomized, double-blind, active-controlled study. Initially, patients will enter a single-blind ramipril run-in period (titrated to 5 mg bid), followed by a sacubitril/valsartan run-in period (100 mg titrated to 200 mg bid). A total of 666 patients tolerating both periods will be randomized 1:1 to either ramipril 10 mg bid or sacubitril/valsartan 200 mg bid. The primary endpoint will be the change of left ventricular end-systolic volume index within 12-month of treatment as measured by magnetic resonance imaging. The main secondary endpoints include the change of left ventricular end-diastolic volume index within 12-month of treatment, the change of LVEF within 12-month of treatment, 12-month composite endpoint of cardiovascular death or heart failure requiring hospitalization, 12-month cardiovascular death, 12-month heart failure requiring hospitalization, time to death or heart failure requiring hospitalization or mortality rate within 12-month of treatment.

This study may determine the place of sacubitril/valsartan as an alternative to ramipril in the treatment of patients with ischemic HFmrEF in order to prevent further left ventricular remodeling and to improve its systolic function.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study, expressed prior to any procedures related to the study.
* Age 18 and over.
* Symptomatic HF in NYHA class II to IV of ischemic etiology.
* Left ventricular ejection fraction at screening visit ranged from 40-49%.
* Elevated concentration of NT-proBNP natriuretic peptide ≥125 pg/ml.
* Features of a structural / functional disease of the left ventricle.
* Optimal pharmacotherapy with ACEI or ARB and beta-blocker, unless they are contraindicated.

Exclusion Criteria:

* History of hypersensitivity or allergy to any of the drugs tested or drugs of similar chemical class, ACEIs, ARBs or neprilysin inhibitors.
* Previous history of intolerance to recommended ACEI or ARB target doses.
* Known history of angioedema.
* Requirement of simultaneous treatment with ACEI and ARB.
* Acute decompensated HF within 6 weeks prior to screening visit.
* Symptomatic hypotension systolic blood pressure <100 mmHg at screening visit.
* Current or previous treatment with sacubitril / valsartan.
* Estimated creatinine clearance <30 ml / min / 1.73 m2 at screening visit.
* Serum potassium >5.2 mmol / L at screening visit.
* Acute coronary syndrome or elective revascularization within 6 weeks prior to screening.
* Stroke, transient ischemic attack, carotid angioplasty, heart surgery, or any other major cardiovascular surgery in the 3 months prior to screening.
* Implantation of a cardioverter defibrillator, pacemaker, or resynchronization therapy device incompatible with MRI.
* Fixed atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular end-systolic volume | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the change in left ventricular end-systolic volume as measured by MRI in patients with ischemic HFmrEF

SECONDARY OUTCOMES:
Change in left ventricular end-diastolic volume | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the change in left ventricular end-diastolic volume as measured by MRI in patients with ischemic HFmrEF
Change in indexed left ventricular end-systolic and end-diastolic volumes | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the change in indexed left ventricular end-systolic and end-diastolic volumes as measured by MRI in patients with ischemic HFmrEF
Change in left ventricular ejection fraction | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the change in left ventricular ejection fraction as measured by MRI in patients with ischemic HFmrEF
Occurrence of the endpoint of death from cardiovascular causes or first hospitalization for HF | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of the endpoint of death from cardiovascular causes or first hospitalization for HF in patients with ischemic HFmrEF
Occurrence of the endpoint of death from cardiovascular causes or first or subsequent hospitalization for HF | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of the endpoint of death from cardiovascular causes or first or subsequent hospitalization for HF in patients with ischemic HFmrEF
Occurrence of death from cardiovascular causes | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of death from cardiovascular causes in patients with ischemic HFmrEF
First hospitalization due to HF | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the first hospitalization due to HF in patients with ischemic HFmrEF
Occurrence of the first or subsequent hospitalization due to HF | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of the first or subsequent hospitalization due to HF in patients with ischemic HFmrEF
Time to death from cardiovascular causes or first hospitalization for HF | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the time to death from cardiovascular causes or first hospitalization for HF in patients with ischemic HFmrEF
Occurrence of death from any cause | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of death from any cause in patients with ischemic HFmrEF

OTHER OUTCOMES:
Incidence of hypotension | 12 months
  Incidence of symptomatic hypotension and/or hypotension with systolic blood pressure <95 mmHg in patients on sacubitril / valsartan versus in those on ramipril
Occurrence of hyperkalaemia | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the occurrence of hyperkalaemia (>5.4 mmol/L)
Onset or worsening of renal failure | 12 months
  Assessment of the effect of sacubitril / valsartan versus ramipril on the onset or worsening of renal failure (eGFR <30 ml / minute / 1.73 m2 or decrease in eGFR compared to visit W1 or W2 by more than 25%)

CONTACTS AND LOCATIONS:
Locations (1):
- Krakowski Szpital Specjalistyczny im. św. Jana Pawła II, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No